CLINICAL TRIAL: NCT03519867
Title: A Multi-center, Randomized, Assessor-blinded, Phase II, Parallel Dose-finding Trial in Subjects of ASA Class 1 - 3 to Assess the Efficacy and Safety of 5 Doses of Org 25969 When Administered at 1-2 PTCs After Administration of Zemuron®
Brief Title: Efficacy and Safety of Org 25969 Administered After Zemuron® (MK-8616-042)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06387; MK-8616-042 (Other: Merck Protocol Number); 19.4.204 (Other: Organon Protocol Number)
Record Dates: First submitted 2018-05-08; First posted 2018-05-09 (Actual); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 0.5 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced neuromuscular blockade (NMB) reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 2) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 0.5 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 3) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 1.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 4) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 1.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 5) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 2.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 6) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 2.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 7) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 4.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 8) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 4.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 9) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 8.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®
- 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg (Experimental): Participants (ASA Class 1 to 3) will receive an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 8.0 mg/kg iv during a single study session. MK-8616 will be administered once Zemuron®-induced NMB reaches 1 to 2 PTCs.
  Interventions: Drug: MK-8616; Drug: Zemuron®

INTERVENTIONS:
Drug: MK-8616 — MK-8616 will be administered at doses of 0.5, 1.0, 2.0, 4.0 and 8.0 mg/kg iv as a 30-second infusion. Doses are based on actual body weight.
  Other Names: Org 25969, sugammadex, Bridion®
Drug: Zemuron® — Zemuron® (0.6 or 1.2 mg/kg, iv) will be administered as a 10-second bolus infusion to achieve 1 to 2 PTCs. If needed, a maintenance dose of 0.15 mg/kg will be given. Doses are based on actual body weight.
  Other Names: Rocuronium bromide

SUMMARY:
The primary objective of this study is to explore the dose-response relation of MK-8616 (Org 25969) given as a reversal agent of Zemuron® at 1 to 2 post tetanic counts (PTCs); both Zemuron® and MK-8616 are administered by intravenous (iv) infusion. Another goal of the study is to evaluate the safety of single doses of MK-8616 administered to participants of American Society of Anesthesiologists (ASA) Physical Status Class 1 (otherwise normal, healthy participant); Class 2 (participant with a mild systemic disease); or Class 3 (participant with a severe systemic disease that limits activity, but is not incapacitating).

ELIGIBILITY:
Inclusion Criteria:

* Has an ASA Class of 1 to 3
* Is scheduled for surgical procedures (excluding dental and neck surgeries) with an anticipated duration of anesthesia of ≥45 minutes with the use of Zemuron®

Exclusion Criteria:

* Is undergoing dental or neck surgery
* Has anatomical malformation that would impede intubation
* Has or is suspected to have neuromuscular disorders impairing neuromuscular block and/or significant renal dysfunction
* Is known or suspected to have a family history of malignant hyperthermia
* Is known or suspected to have an allergy to narcotics, muscle relaxants, or other medications used during general anesthesia
* Is pregnant
* Is a female of childbearing potential not using 1 of the following methods of birth control: condom or diaphragm with spermicide, vasectomized partner (<6 months), intrauterine device (IUD), or abstinence
* Is breast-feeding
* Has already participated in the study
* Has participated in another clinical trial, not pre-approved by Organon Pharmaceuticals USA within 30 days of entering this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2005-05-26 (Actual); Study Completion 2005-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants of American Society of Anesthesiologists (ASA) Class 1-3 who were scheduled for surgery were recruited at 4 study sites in the US.
Groups:
- 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 0.5 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced neuromuscular blockade (NMB) reached 1 to 2 PTCs.
- 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 1.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 2.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 4.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 8.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 0.5 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 1.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 2.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 4.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 1.2 mg/kg followed by MK-8616 8.0 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
Period: Overall Study
Arm/Group | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg
Started | 6 | 7 (One participant randomized to receive MK-8616 8.0 mg/kg received MK-8616 0.8 mg/kg.) | 6 | 4 | 5 | 5 | 4 | 5 | 4 | 4
Treated | 5 | 6 | 5 | 3 | 5 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 5 | 3 | 5 | 2 | 3 | 4 | 3 | 4
Not Completed | 3 | 3 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Admin. of relaxant other than Zemuron® | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Admin. of other reversal agent | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Reason not provided | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for all treated participants.
Groups:
- 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg: Participants (ASA Class 1 to 3) received an iv bolus of Zemuron® 0.6 mg/kg followed by MK-8616 0.5 mg/kg iv during a single study session. MK-8616 was administered once Zemuron®-induced NMB reached 1 to 2 PTCs.
- Total: Total of all reporting groups
Arm/Group | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg | Total
Number analyzed (Participants) | 5 | 6 | 5 | 3 | 5 | 4 | 4 | 4 | 3 | 4 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All treated participants.
  Years | 48 (12) | 49 (10) | 52 (11) | 58 (20) | 53 (14) | 58 (11) | 47 (12) | 51 (4) | 48 (17) | 50 (10) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants.
  Participants
    Female | 2 | 3 | 2 | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 21
    Male | 3 | 3 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of MK-8616 to Recovery T4/T1 Ratio to 0.9
Description: The mean time from the start of MK-8616 administration to recovery T4/T1 ratio of 0.9 was determined. Less time indicates faster recovery from NMB. The ratio of T4 (fourth twitch; amplitude of fourth response to train of four [TOF] stimulation is expressed as percent of control T4) over T1 (first twitch; amplitude of first response to TOF stimulation is expressed as percent of control T1) ranges from 0 (complete loss of T4 twitch response) to 1.0 (complete recovery of T4 twitch response). For TOF stimulation, 4 consecutive square wave supra-maximal stimuli of 0.2 msec duration were delivered at 2 Hz every 15 seconds. Neuromuscular monitoring was performed with the TOF-Watch® SX.
Time Frame: Up to 90 minutes
Population: All randomized participants who received ≥1 dose of study drug, had ≥1 post baseline efficacy measurement, and did not have any important protocol violations are included.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg
Number analyzed (Participants) | 3 | 2 | 5 | 2 | 4 | 1 | 3 | 3 | 2 | 4
Minutes | 44.18 (34.63) | 19.08 (19.98) | 5.38 (5.57) | 3.32 (1.63) | 1.53 (0.60) | 20.57 (0) | 11.52 (11.63) | 4.33 (0.52) | 1.92 (0.65) | 0.98 (0.18)

2. Secondary Outcome: Percentage of Participants Experiencing ≥1 Adverse Events (AEs)
Description: The percentage of participants experiencing ≥1 AEs was determined. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 7 days following MK-8616 administration
Population: All participants who received a dose of study treatment are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg
Number analyzed (Participants) | 5 | 6 | 5 | 3 | 5 | 4 | 4 | 4 | 3 | 4
Percentage of Participants | 100.0 | 100.0 | 60.0 | 66.7 | 80.0 | 100.0 | 100.0 | 100.0 | 66.7 | 50.0

ADVERSE EVENTS:
Time Frame: Up to 7 days
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. All participants who received a dose of study treatment are included.
Arm/Group | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/3 | 0/5 | 0/4 | 0/4 | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 0/5 | 1/3 | 1/5 | 0/4 | 0/4 | 1/4 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 3/5 | 1/3 | 4/5 | 4/4 | 4/4 | 4/4 | 2/3 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg (N=5) | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg (N=6) | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg (N=5) | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg (N=3) | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg (N=5) | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg (N=4) | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg (N=4) | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg (N=4) | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg (N=3) | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg (N=4)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1) Zemuron® 0.6 mg/kg + MK-8616 0.5 mg/kg (N=5) | 2) Zemuron® 0.6 mg/kg + MK-8616 1.0 mg/kg (N=6) | 3) Zemuron® 0.6 mg/kg + MK-8616 2.0 mg/kg (N=5) | 4) Zemuron® 0.6 mg/kg + MK-8616 4.0 mg/kg (N=3) | 5) Zemuron® 0.6 mg/kg + MK-8616 8.0 mg/kg (N=5) | 6) Zemuron® 1.2 mg/kg + MK-8616 0.5 mg/kg (N=4) | 7) Zemuron® 1.2 mg/kg + MK-8616 1.0 mg/kg (N=4) | 8) Zemuron® 1.2 mg/kg + MK-8616 2.0 mg/kg (N=4) | 9) Zemuron® 1.2 mg/kg + MK-8616 4.0 mg/kg (N=3) | 10) Zemuron® 1.2 mg/kg + MK-8616 8.0 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 2 (3) | 1 (1) | 2 (2)
Post procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuromuscular blockade (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Organon recognizes the right of the investigator(s) to publish, but all publications must be based on data validated by Organon. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to Organon, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.